CLINICAL TRIAL: NCT05985460
Title: A Very Brief Intervention to Increase the Intention to Practice Physical Activity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JCSFLP2
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Physical Activity
Keywords: Family Well-being; Physical Activity; Health; Digital Game
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: motion-sensor video game (Experimental): The experimental arm is a 1-2 mins motion-sensoring video game, which can accommodate 1-4 individuals, engaging their entire bodies in the physical motions involved. It aims to increase PA intention by increasing their motivation, as well as personal and family well-being by increasing the interaction with family members. Assessments will be conducted at two different time points, immediately following the intervention (T2) and after 1-month follow-up (T3).
  Interventions: Device: Intervention: motion-sensor video game
- Placebo: mobile APP game (without motion-sensoring) (Placebo Comparator): The placebo arm is a 1-2 mins mobile app game, which allows 1-4 participants to play together with a duration of 1-2 minutes. It aims to increase participants' family and personal well-being by increasing the interaction of family members. Assessments will be conducted at two different time points, immediately following the intervention (T2) and after 1-month follow-up (T3).
  Interventions: Device: Placebo: mobile APP game (without motion-sensoring)

INTERVENTIONS:
Device: Intervention: motion-sensor video game — The experimental arm is a 1-2 mins motion-sensoring video game, which can accommodate 1-4 individuals, engaging their entire bodies in the physical motions involved. It aims to increase PA intention by increasing their motivation, as well as personal and family well-being by increasing the interaction with family members. Assessments will be conducted at two different time points, immediately following the intervention (T2) and after 1-month follow-up (T3).
  Arms: Intervention: motion-sensor video game
Device: Placebo: mobile APP game (without motion-sensoring) — The placebo arm is a 1-2 mins mobile app game, which allows 1-4 participants to play together with a duration of 1-2 minutes. It aims to increase participants' family and personal well-being by increasing the interaction of family members. Assessments will be conducted at two different time points, immediately following the intervention (T2) and after 1-month follow-up (T3).
  Arms: Placebo: mobile APP game (without motion-sensoring)

SUMMARY:
According to the Health Belief Model (HBM), one's intention to engage in physical activity (PA) is strongly and favourably related to their actual PA behaviour (Etheridge, Sinyard, & Brindle, 2023; Kagee & Freeman, 2017). According to a meta-analysis that looked at the connection between PA intention and conduct, 54% of those who had the intention to be active did so, and just 2% of people who initially had no intention of engaging in PA later modified their behaviour (Rhodes & de Bruijn, 2013). Therefore, having PA intention is a crucial and helpful step to participate in PA(Webb & Sheeran, 2006).

Digital games include TV or console games, PC games, portable games, and others. Such games have recently been employed as teaching, learning, and training aids in a variety of contexts, including medical education (Rosenberg et al., 2010). Previous research has shown that motion sensor video games have positive effects on promoting healthy lifestyles including engagement in physical activity and disseminating health-related knowledge (DeSmet et al., 2014; Foley & Maddison, 2010; Lenhart, Kahne, Middaugh, Evans, & Vitek, 2008). Meanwhile, video games (at least once/day for 1 week) had positive effects on individuals' well-being and family relationships. (Foley & Maddison, 2010; Halbrook, O'Donnell, & Msetfi, 2019). Drawing on the HBM, playing digital game could be the cue to action which increases people's intention to engage in physical activities.

Our study aims to fill the gap by examining the effectiveness of motion-sensoring game-based intervention in increasing the intention of performing PA, as well as personal and family well-being.

DETAILED DESCRIPTION:
Health promotion refers to the process through which individuals are empowered to enhance their control over their health and work towards its improvement (Smith, Tang, & Nutbeam, 2006). The primary obstacles encountered in prior health promotion initiatives predominantly involve participant engagement and the allocation of adequate resources for execution (Korda, 2013). Owing to the rapid digital transformation in recent decades, digital games are becoming increasingly popular approaches for health promotion that could cover the above challenges.

Regular physical activity is proven to help prevent and manage noncommunicable diseases (NCDs) such as heart disease, stroke, diabetes and several cancers. It also helps prevent hypertension, maintain healthy body weight and can improve mental health, quality of life and well-being. Intention is such a strong psychological predictor of behaviour including PA, as a result, PA intention has been an important and useful precursor to PA participation.

Therefore, our study aims to explore the effectiveness of motion-sensoring game-based intervention in increasing intention to perform physical activity. The intervention is a kind of motion-sensoring game based on Nintendo Switch that can accommodate 1-4 individuals, engaging their entire bodies in the physical motions involved and will last 1-2 minutes each session. It is notable that our project apps, a kind of mobile game, will be a placebo that was developed to promote family well-being in Hong Kong, has been applied in previous community events and received high satisfaction and positive feedback from both community participants and NGO social workers. We hypothesize that the motion-sensoring would promote the intention on participating in PA, as well as self-perceived personal and family well-being.

The primary objective is to promote the intention to perform physical activity. The secondary objectives are to enhance the knowledge of PA and to enhance their personal and family well-being.

ELIGIBILITY:
Inclusion Criteria:

* Chinese speaking
* Able to complete the questionnaire
* Aged 18 or above

Exclusion Criteria:

* People with serious health conditions that might prevent them from participating in sensor-motion video game and mobile game

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2023-09-05 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Intention to perform physical activity | Immediate post-intervention, 1-month follow up
  The intention to perform physical activity will be assessed immediately following the activity and after 1-month follow-up by one-item scale. The question is "Do you want to start (or continue) exercising at present?". The item comprises a 11-point scale ranging from 0 to 10 (Lin, Huang, Chuang, Tsai, & Wang, 2018).

SECONDARY OUTCOMES:
Satisfaction with the games • personal well-being and family well-being | Immediate post-intervention, 1-month follow up
  The question "Are you satisfied with this activity?" will be used to assess the satisfaction of participants after playing the two kinds of games and 1-month follow-up with a higher score (1-5) indicating higher satisfaction.
Personal well-being and family well-being | Immediate post-intervention, 1-month follow up
  Personal well-being was assessed immediately after playing games and 1-month follow-up using the question "How well-being do you think you are?" and answer using the 11-point scale (range 0-10), with higher scores indicating higher level of family well-being. (Appendix H1, H2) Family well-being was measured immediately after playing games and 1-month follow-up using family health, harmony, and happiness (3Hs): three separate questions asked, "How healthy/harmonious/happy do you think your family is?" and were answered using an 11-point scale ranging from 0 to 10, with higher scores indicating higher level of family well-being. (Appendix H1, H2)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeSmet A, Van Ryckeghem D, Compernolle S, Baranowski T, Thompson D, Crombez G, Poels K, Van Lippevelde W, Bastiaensens S, Van Cleemput K, Vandebosch H, De Bourdeaudhuij I. A meta-analysis of serious digital games for healthy lifestyle promotion. Prev Med. 2014 Dec;69:95-107. doi: 10.1016/j.ypmed.2014.08.026. Epub 2014 Aug 27. PMID 25172024
- [Background] Etheridge, J. C., Sinyard, R. D., & Brindle, M. E. (2023). Chapter 90 - Implementation research. In A. E. M. Eltorai, J. A. Bakal, P. C. Newell, & A. J. Osband (Eds.), Translational Surgery (pp. 563-573): Academic Press.
- [Background] Foley L, Maddison R. Use of active video games to increase physical activity in children: a (virtual) reality? Pediatr Exerc Sci. 2010 Feb;22(1):7-20. doi: 10.1123/pes.22.1.7. PMID 20332536
- [Background] Halbrook YJ, O'Donnell AT, Msetfi RM. When and How Video Games Can Be Good: A Review of the Positive Effects of Video Games on Well-Being. Perspect Psychol Sci. 2019 Nov;14(6):1096-1104. doi: 10.1177/1745691619863807. PMID 31672105
- [Background] Kagee, A., & Freeman, M. (2017). Mental Health and Physical Health (Including HIV/AIDS). In S. R. Quah (Ed.), International Encyclopedia of Public Health (Second Edition) (pp. 35-44). Oxford: Academic Press.
- [Background] Korda H. Bringing evidence-based interventions to the field: the fidelity challenge. J Public Health Manag Pract. 2013 Jan-Feb;19(1):1-3. doi: 10.1097/PHH.0b013e318249bc06. PMID 23169396
- [Background] Lenhart, A., Kahne, J., Middaugh, E., Evans, C., & Vitek, J. (2008). Teens' gaming experiences are diverse and include significant social interaction and civic engagement. Pew Internet and American Life Project. Retrieved April 2, 2009. In.
- [Background] Lin ML, Huang JJ, Chuang HY, Tsai HM, Wang HH. Physical activities and influencing factors among public health nurses: a cross-sectional study. BMJ Open. 2018 Apr 20;8(4):e019959. doi: 10.1136/bmjopen-2017-019959. PMID 29678974
- [Background] Rhodes RE, de Bruijn GJ. How big is the physical activity intention-behaviour gap? A meta-analysis using the action control framework. Br J Health Psychol. 2013 May;18(2):296-309. doi: 10.1111/bjhp.12032. PMID 23480428
- [Background] Rosenberg D, Depp CA, Vahia IV, Reichstadt J, Palmer BW, Kerr J, Norman G, Jeste DV. Exergames for subsyndromal depression in older adults: a pilot study of a novel intervention. Am J Geriatr Psychiatry. 2010 Mar;18(3):221-6. doi: 10.1097/JGP.0b013e3181c534b5. PMID 20173423
- [Background] Smith BJ, Tang KC, Nutbeam D. WHO Health Promotion Glossary: new terms. Health Promot Int. 2006 Dec;21(4):340-5. doi: 10.1093/heapro/dal033. Epub 2006 Sep 7. PMID 16963461
- [Background] Webb TL, Sheeran P. Does changing behavioral intentions engender behavior change? A meta-analysis of the experimental evidence. Psychol Bull. 2006 Mar;132(2):249-68. doi: 10.1037/0033-2909.132.2.249. PMID 16536643